CLINICAL TRIAL: NCT05957315
Title: Mobile Cardiac Outpatient Telemetry for Unexplained Syncope: Time to Treatment, Arrhythmia Diagnosis and Outcome
Brief Title: Mobile Cardiac Outpatient Telemetry for Unexplained Syncope
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Carilion Clinic (Other)
Responsible Party: Principal Investigator, Andrew Moore, Principal Investigator, Carilion Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-22-1733
Record Dates: First submitted 2023-07-14; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Syncope; Arrhythmia; Near Syncope; Arrhythmias, Cardiac
Keywords: Cardiac monitoring; Syncope; Unexplained syncope
MeSH Terms: conditions — Syncope; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Mobile Cardiac Outpatient Telemetry Device (MCOT) (Experimental): These participants will be randomized into receiving the Philips/BioTel MCOT device in addition to usual care.
  Interventions: Device: Mobile Cardiac Outpatient Telemetry Device (MCOT)
- Standard Treatment Group (No Intervention): These participants will be randomized into only receiving usual care and will not receive the MCOT device.

INTERVENTIONS:
Device: Mobile Cardiac Outpatient Telemetry Device (MCOT) — Application of a Philips/Biotel MCOT device
  Other Names: cardiac monitor, cardiac monitoring, mobile cardiac telemetry
  Arms: Mobile Cardiac Outpatient Telemetry Device (MCOT)

SUMMARY:
This study seeks to provide evidence that use of Philips mobile cardiac outpatient telemetry (MCOT) devices may improve patient care for patients who present to emergency departments (EDs) with syncope, which is a temporary loss of consciousness also known as fainting or who present experiencing a near temporary loss of consciousness (near syncope). It is set up as a random controlled trial, which means research participants will be randomly assigned to receiving the device or usual care. Patients 50 years or older who come to the ED of Carilion Roanoke Memorial Hospital will be screened by study team members for unexplained syncope or near syncope across three ED dispositions: hospital admission, emergency department clinical decision unit admission (ED CDU) and emergency department. After consent, subjects will be enrolled and randomized, via REDCap randomization, in the study. At the time of subject discharge the MCOT device will be placed on the chest for the arm of intervention patients (for subjects who were admitted, the research study team will follow the patient's clinical course and placement of the device will occur at discharge); subjects will also receive brief instruction on the care and maintenance of the device and a patient education guide. The research team will contact the subjects for a telephone follow up at 14 and 30 days post-enrollment. The study will establish the efficacy of mobile cardiac outpatient telemetry in comparison to observation telemetry. Research objectives are to 1) Measure the time to medical intervention in patients with unexplained syncope or near syncope fitted with a Philips MCOT at the time of hospital discharge compared to patients treated with usual care for unexplained syncope or near syncope; and 2) Measure the time to arrhythmia diagnosis in patients with unexplained syncope or near syncope fitted with a Philips MCOT at the time of hospital discharge compared to patients treated with usual care for unexplained syncope or near syncope.

DETAILED DESCRIPTION:
The study will establish the efficacy of ED-based, post-discharge mobile cardiac outpatient telemetry for patients discharged with a diagnosis of unexplained syncope.

Research objectives are to 1) Measure the time to medical intervention in patients with unexplained syncope fitted with a Philips MCOT at the time of hospital discharge compared to patients treated with usual care for unexplained syncope; and 2) Measure the time to arrhythmia diagnosis in patients with unexplained syncope fitted with a Philips MCOT at the time of hospital discharge compared to patients treated with usual care for unexplained syncope.

The hypothesis for this study is that participants who receive the Philips MCOT device upon discharge will experience a shorter time to diagnosis for the cause of their episode of syncope and receive subsequent medical intervention sooner than those who do not receive an MCOT device.

Medical intervention is defined as a change in medical management, escalation of diagnostic testing or device, or medical procedure that might result from diagnostic information obtained from outpatient cardiac monitoring following a syncopal episode. Change in medical management includes, but is not limited to, initiation of a new medication, lifestyle modification recommendations, referral to medical specialist such as cardiology or electrophysiology. Escalation of diagnostic device may include, but is not limited to, ordering of diagnostic studies such as a cardiac stress test, echocardiogram, other cardiac testing at the preference of the treating subspecialist, or placement of a longer duration cardiac monitor such as an implantable loop recorder or cardiac event monitor. Medical procedure is defined as cardiac pacemaker implantation, cardiac heart catheterization, or other invasive cardiac procedure felt to be medically necessary by the treating specialist or subspecialist physician.

An arrhythmia is an abnormal heart rhythm. In some instances syncope/near syncope, or fainting/near fainting, may be the result of an undiagnosed abnormal heart rhythm. Abnormal heart rhythms that might result in a fainting include atrial fibrillation, supraventricular tachycardia, sinus pause, Mobitz Type II heart block, complete heart block, and ventricular tachycardia. Wearing the mobile cardiac outpatient telemetry monitor increases the likelihood of identifying fainting episodes that were caused by abnormal heart rhythms.

Previous studies are variable in the number and type of arrythmias captured that would mandate medical intervention of some type that is measurable (medication, ablation, etc). All comer diagnosis and absolute diagnosis of any arrythmia is much higher than 10%. Thus, we based the pilot study size based on the lowest reported incidence in the literature for arrythmias requiring a change in a patient's medical care of 10% as the lowest suspected incidence for the Na sample size calculation. With a one-sided means test, 1-b at 0.80, and a of 0.05, 8 events in Na requiring medical intervention of some type would be required to demonstrate a 7d difference in time to intervention from the usual care group or 80 patients in the Na and 160 total. The device manufacturer is providing up to 120 devices with monitoring (up to 240 total study enrollees), which will allow for flexibility in the event of loss to follow up or to increase power.

Study participants will be randomized at ED discharge into either the control group, which receives usual care (referrals to follow up with outpatient services), or the experimental group, which receives usual care AND are fitted with a Philips MCOT device and remotely monitored for 30 days along with possible referrals to follow up with outpatient services. Data will be collected from participants' medical records to determine whether additional episodes of syncope or near syncope, diagnosis, and/or treatment occurred. Additionally, participants will be contacted by the study team at 14 and 30 days post-discharge to answer questions to determine whether additional episodes of syncope or near syncope occurred, whether treatment occurred, and whether they complied with follow up referrals. To determine if there is a difference in the time to medical intervention and in time to arrhythmia diagnosis, we will conduct two-sample tests of proportions. Secondary outcome analysis will be descriptive.

ELIGIBILITY:
Inclusion Criteria:

ED presentation for syncope or near syncope without identified cause of syncope during ED evaluation

Willingness to enroll in the trial

greater than or equal to 50 years of age

cell phone coverage at their primary residence

home or cell phone service for follow up calls

ability to answer questionnaires without assistance

English language speaker

Exclusion Criteria:

unwillingness to participate in the study

unable to consent on their own

seizure as presumptive cause of loss of consciousness

stroke, or transient ischemic attack as presumptive loss of consciousness

loss of consciousness following head trauma

confusion from baseline mental status (altered mental status)

intoxication (alcohol or other drugs)

medical or electrical intervention required to restore consciousness

hypoglycemia as presumptive cause of loss of consciousness

inability to provide follow up via telephone (phone that is not regularly in service)

lack of permanent address (e.g. not a homeless shelter, half-way house, psychiatric treatment facility, or correctional facility)

Lack of continuous cellular phone service with ATT, Verizon, or T-Mobile for MCOT relay

known pregnancy

Illiteracy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Time to arrhythmia diagnosis for unexplained syncope | 1 month
  Comparison of time to arrhythmia diagnosis for intervention vs. control group
Time to medical intervention following unexplained syncope | 1 month
  Comparison of time to medical intervention for intervention vs. control group